CLINICAL TRIAL: NCT00826696
Title: A Retrospective Review of the Seasonality of Pre-Eclampsia
Status: Completed | Type: Observational
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Nicole Bullock, D.O., OSUCHS Department of Obstetrics and Gynecology
Other Study IDs: 2008021
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Preeclampsia
Keywords: preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This retrospective review will will attempt to determine whether our data show a significant difference in number of deliveries of women with pre-eclampsia compared to deliveries without pre-eclampsia during certain months of the year.

DETAILED DESCRIPTION:
This study is a retrospective review of obstetrics charts of women who gave birth at OSU Medical Center between January 01, 2005 and December 31, 2007.

Included will be patient charts of women > 18 years old who were admitted to OSUMC for delivery (both cesarean and vaginal deliveries) between 1/1/05 and 12/31/07, with and without a diagnosis of pre-eclampsia. The data collected will be recorded in a spreadsheet by month/day of delivery, and whether pre-eclampsia was a diagnosis. Also included will be total number of deliveries per month and total number of pre-eclampsia diagnoses per month. The rate of pre-eclampsia will be calculated.

A contingency table with corresponding chi square test will be performed to determine whether there is a significant relationship of the diagnosis of pre-eclampsia with seasonality, defined primarily by month. Certain data occurring during transition periods between seasons may be excluded from analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth at OSU Medical Center between January 01, 2005 and December 31, 2007 and were > 18 years old who were admitted to OSUMC for delivery (both cesarean and vaginal deliveries) between 1/1/05 and 12/31/07, with and without a diagnosis of pre-eclampsia.

Exclusion Criteria:

* Females under age 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women of all races who were admitted to OSUMC for delivery of a baby (both cesarean and vaginal deliveries) between 1/1/05 and 12/31/07, with or without a diagnosis of pre-eclampsia.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of women per month who had a diagnosis of pre-eclampsia at OSU Medical Center when they delivered a baby. | Data assessed from patient charts retrospectively

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bullock, DO, Principal Investigator — OSU Center for Health Sciences
Locations (1):
- Oklahoma State University Medical Center, Tulsa, Oklahoma, United States